CLINICAL TRIAL: NCT02636803
Title: An Open Comparative Study of the Efficacy of Different Doses of Oxfendazole Compared to Single Dose Albendazole in the Treatment of Trichuris Trichiura Infection in Adults
Brief Title: Study of the Efficacy of Oxfendazole Compared to Albendazole in the Treatment of Trichuris Trichiura Infection in Adults
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: not going to be conducted
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Universidad Peruana Cayetano Heredia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: OXF2
Record Dates: First submitted 2015-12-14; First posted 2015-12-22 (Estimated); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Helminthiasis
Keywords: trichuris; hookworms; Ascaris
MeSH Terms: conditions — Helminthiasis; Hookworm Infections | interventions — oxfendazole; Albendazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- oxfendazole 6 mg/kg (Experimental): patients receive 6 mg/kg oxfendazole once
  Interventions: Drug: oxfendazole
- oxfendazole 30 mg/kg (Experimental): patients receive 30 mg/kg oxfendazole once
  Interventions: Drug: oxfendazole
- oxfendazole 6 mg/kg 3 times (Experimental): patients receive 6 mg/kg oxfendazole three times
  Interventions: Drug: oxfendazole
- albendazole 400 mg (Active Comparator): patients receive 400 mg albendazole once
  Interventions: Drug: albendazole

INTERVENTIONS:
Drug: oxfendazole — group receives a single dose of oxfendazole at 6 or 30 mg/kg or three 6 mg/kg doses
  Arms: oxfendazole 30 mg/kg; oxfendazole 6 mg/kg; oxfendazole 6 mg/kg 3 times
Drug: albendazole — group receives one 400 mg dose of albendazole
  Arms: albendazole 400 mg

SUMMARY:
The aim of this study is to provide data on the efficacy of oxfendazole against Trichuris trichiura at different doses in comparison to the standard single 400 mg dose of albendazole. In addition, the study will provide data on oxfendazole efficacy against other common nematodes encountered in man (Enterobius vermicularis, Ascaris lumbricoides, Ancylostoma duodenalis, Necator americanus).

DETAILED DESCRIPTION:
This is an open, comparative study in adult patients with proven intestinal infection with Trichuris trichiura. Patients meeting the study entry criteria will receive either 6mg/kg, or 30 mg/kg of oxfendazole as a single oral dose or 6 mg/kg orally for three days or albendazole 400mg as a single oral dose. Stool samples will be obtained and examined 7, 14 and 21 days after treatment.

Two hundred clinically evaluable patients of either gender, 16 - 65 years of age, presenting with proven Trichuris trichiura infection, recruited from one centre, will be included in the study. there will be 15 patients in each treatment group. Duration of accrual will be determined in discussion with the clinical site in Iquitos, Peru.

ELIGIBILITY:
Inclusion Criteria:

1. Written or witnessed oral informed consent has been obtained.
2. Has Trichuris trichiura demonstrated in stool samples obtained during the week before enrolment: The presence of other helminths: Enterobius vermicularis, Ascaris lumbricoides, Necator americanus, Ancylostoma duodenalis will not be a cause for exclusion.
3. Is willing to comply with the requirements of the protocol and particularly to provide 4 stool samples, pretreatment and 7, 14 and 21 days after treatment.
4. Female patients of child bearing potential, who are using an established method of birth control (surgically sterile, intra-uterine contraceptive device, oral contraceptives, diaphragm in combination with contraceptive cream or foam, or condom in combination with contraceptive cream or foam)

Exclusion Criteria:

1. The patient has demonstrated a previous hypersensitivity reaction to benzimidazole or other related compound.
2. Presence of other helminths without Trichuris trichiura. Note: Non-target species may be present and details of response will be recorded.
3. The patient has diarrhoeal disease that would interfere with the evaluation of stool samples.
4. The patient has received an anthelminthic in the 2 weeks prior to enrolment into the study.
5. The patient has received an investigational drug within 30 days or 5 half-lives (whichever is longer) of the screening visit or is scheduled to receive such a drug during the study period.
6. The patient has a concomitant infection or any other underlying disease that would compromise the diagnosis and the evaluation of the response to the study medication.
7. The patient has a known history of renal dysfunction (plasma creatinine ≥ 1.5 times upper limit of normal for age) or hepatic dysfunction (liver enzymes ≥ 1.5
8. Is a female who is pregnant, lactating or planning a pregnancy during the study, or is not practicing any form of contraception (see inclusion criteria (4.2.5).
9. Patient that is unwilling or unable to take part in this study.
10. The patient has previously been enrolled in the study.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
Cure of Trichuris trichiura | day 21 following treatment
  Cure of infection (Clinical Cure) shown by absence of Trichuris eggs in stool examinations at Day 21, using Kato Katz test.
Reduction in Trichuis trichiura eggs (compared to pretreatment) | day 21 following treatment
  Reduction (compared to baseline) of Trichuris eggs in stool examinations at 21, using Kato Katz test.

SECONDARY OUTCOMES:
Cure of other intestinal helminths | day 21 following treatment
  Absence of Ascaris, Necator eggs in stool using Kato Katz test
Safety and tolerability of oxfendazole in the treatment of adult patients assessed by cumulative adverse events | treatment through day 21 following treatment
  Cumulative adverse events following treatment up to Day 21

CONTACTS AND LOCATIONS:
Overall Officials: Robert H Gilman, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Hector H Garcia, MD, PhD, Principal Investigator — Universidad Peruana Cayetano Heredia; Richard J Horton, MB BChir, MRCGP, FFPM, Principal Investigator — Tropical Projects; Armando E Gonzalez, DVM, PhD, Principal Investigator — National University of San Marcos, Peru

IPD SHARING:
Plan to Share IPD: Yes
posting to CT.gov and publication